CLINICAL TRIAL: NCT03055299
Title: Comprehensive Exercise (COMEX) Program for Dialysis Patients Pilot Study
Brief Title: COMEX Study for Dialysis Patients
Acronym: COMEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Manisha Jhamb, MD, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO15070086
Record Dates: First submitted 2017-01-23; First posted 2017-02-16 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COMEX (Experimental): Patients receive comprehensive exercise intervention
  Interventions: Other: COMEX intervention

INTERVENTIONS:
Other: COMEX intervention — Comprehensive Exercise

SUMMARY:
The goal of the COMprehensive EXercise (COMEX) pilot study is to test feasibility, tolerability and adherence of this novel video-based intra-dialytic chair exercise program for hemodialysis patients over 3 months.

DETAILED DESCRIPTION:
The investigators incorporated patient-provider preferences of the key stakeholders, and used a multi-disciplinary team with experts in physical therapy, psychology and nephrology to develop a comprehensive exercise program for HD patients. Aim of this pilot study is to assess the feasibility, tolerability and adherence to COMEX over 3 months and inform design of future randomized controlled trial. A secondary goal is to explore molecular mechanisms in muscle and blood of exercise adaptation in HD patients

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Age ≥18 years to 85 years
* Undergoing maintenance hemodialysis for >3 months at one of the participating dialysis sites
* Patients must be willing and able to sign the consent form.

For providers:

* Eligible if they are a registered nurse, dialysis technician, dialysis social worker, dietitian, dialysis unit administrator or nephrologist involved in providing care for one of the patient participants in the study

Exclusion Criteria:

For all patients:

* Uncontrolled BP (>180/100 mm Hg)
* Inadequately dialyzed (Kt/V<1.2)
* History of Intradialytic hypotension (SBP<90mm Hg) or hypertension (SBP>180mmHg) during/post dialysis within last 1 month
* Contraindication to exercise eg unstable angina, uncompensated congestive heart failure
* Refractory/untreated psychiatric disorders
* History of poor adherence to HD treatment.
* Scheduled for living donor kidney transplant, intention to change to peritoneal dialysis, home HD, or plans to relocate to another center within the next 6 months.
* Currently in acute or chronic care hospital
* Life expectancy < 6 months or intention to withdraw dialysis therapy within 6 months.
* Current pregnancy, or actively planning to become pregnant in the next 6 months
* Currently a prisoner
* Current use of investigational drugs or participation in another non-observational clinical trial that contradicts or interferes with the therapies or measured outcomes in this trial
* Unable or unwilling to follow the study protocol for any reason (including mental incompetence)
* Unable or unwilling to provide informed consent or sign IRB-approved consent form
* Has a tunneled dialysis catheter
* If diabetic, blood sugar control is not stable

For patients undergoing biopsy and blood draw:

* Allergy to lidocaine
* Anemia, <10.0 Hgb
* Chronic use of oral corticosteroids or other medication that affect muscle function
* Any bleeding disorder that would contraindicate biopsy or blood draw such as a history of clinically significant bleeding diathesis (e.g. hemophilia A or B, Von Willebrand's Disease or congenital Factor VII deficiency)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 3 months
  Feasibility will be estimated by calculating the % of eligible participants who consent to participate in the study.
Number of participants with exercise-related adverse events | 3 months
  Tolerability will be measured by assessing exercise related side effects - this will be done by weekly patient interviews and review of medical records
Adherence rate | 3 months
  Adherence will be calculated as % of participants who complete the 3 month COMEX intervention. Also, adherence to exercise will be calculated as % of exercise sessions completed

SECONDARY OUTCOMES:
Fatigue | 3 months
  Self reported fatigue using Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Fatigue questionnaire will be measured at baseline and at 3 months
Sleep | 3 months
  Self reported sleep using Pittsburgh Sleep Quality Index (PSQI) questionnaire will be measured at baseline and at 3 months
Depression | 3 months
  Self reported depression using Beck's Depression Inventory -II questionnaire will be measured at baseline and at 3 months
Global health | 3 months
  Self reported HRQOL using NIH Patient Reported Outcomes Measurement Information System (PROMIS) Adult Global Health questionnaire will be measured at baseline and at 3 months
Health related quality of life | 3 months
  Self reported HRQOL using Short-Form 36 questionnaire will be measured at baseline and at 3 months
Sleep/Wake Behavior by Actigraphy | 3 months
  Objective sleep and activity will be measured using actigraphy
Physical functioning | 3 months
  Will be measured by Short Physical Performance battery at baseline and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Jhamb M, Devaraj SM, Alemairi M, Lavenburg LM, Shiva S, Yabes JG, Forman DE, Hergenroeder AL. A Comprehensive Exercise (COMEX) Intervention to Optimize Exercise Participation for Improving Patient-Centered Outcomes and Physical Functioning in Patients Receiving Hemodialysis: Development and Pilot Testing. Kidney Med. 2023 Sep 12;5(11):100720. doi: 10.1016/j.xkme.2023.100720. eCollection 2023 Nov. PMID 37928754